CLINICAL TRIAL: NCT01265277
Title: Changes in Sleep Patterns and Stress in Infants Entering Child Care: Implications for SIDS Risk
Brief Title: Changes in Sleep Patterns and Stress in Infants Entering Child Care
Status: Completed | Type: Observational
Sponsor: Rachel Moon, MD (Other)
Responsible Party: Sponsor-Investigator, Rachel Moon, MD, MD, University of Virginia
Organization: University of Virginia (Other)
Other Study IDs: 4453
Record Dates: First submitted 2010-12-20; First posted 2010-12-23 (Estimated); Last update posted 2018-12-10 (Actual); Status verified 2018-12

CONDITIONS: Sudden Infant Death Syndrome
Keywords: sudden infant death syndrome; SIDS; infant; licensed day care; sleep patterns; stress levels
MeSH Terms: conditions — Sudden Infant Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — urine samples from both mom and baby
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- at home: Infants 0-3 months who will stay at home with a parent
- child care: Infant 0-3 months who will attend a licensed child care center

SUMMARY:
When babies start day care, they experience many changes, some of which may affect their risk for sudden infant death syndrome (SIDS). The investigators want to find out if stress or change in the baby's sleep patterns can be a reason for this increased risk for SIDS.

DETAILED DESCRIPTION:
The overall aim of this study is to describe sleep patterns in infants as they transition from home to child care, including 24-hour sleep duration, changes in the timing of daytime naps, and changes in nocturnal sleep periods; to describe potential sleep disrupters, such as temperature, light and noise, in home and child care settings that may impact sleep quality and sleep patterns; to describe markers of parent and infant stress levels during the transition to child care; to describe markers of infant circadian rhythm during the transition to child care.

ELIGIBILITY:
Inclusion Criteria:

* Infants who are less than 3 months of age from English-speaking families where one or both parents live in the household will be eligible to participate. If the infant will be entering child care, the infant must be entering a licensed child care center, and child care entry must be between 60 and 120 days of age.

Exclusion Criteria:

* S/he was born prematurely, with a gestational age less than 37 weeks at birth, or had a birth weight <2500 grams (5-1/2 lbs)
* S/he has any medical problems that require ongoing care by a subspecialty physician

Max Age: 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: infants from 0 to 3 months in the United States
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2009-07 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Sleep efficiency | Days -14 through +14
  sleep efficieny is defined as the ratio of time spent asleep (total sleep time) to the amount of time spent in bed.

SECONDARY OUTCOMES:
Sleep duration | Days -14 to +14

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Y Moon, MD, Principal Investigator — University of Virginia
Locations (1):
- Children's National Medical Center, Washington D.C., District of Columbia, United States